CLINICAL TRIAL: NCT07214766
Title: A Phase 1, Randomized, Two-Part, Parallel-Group Study to Assess the Bioequivalence of Subcutaneously Administered Trastuzumab Via Different Subcutaneous Delivery Platforms in Healthy Male Subjects
Brief Title: A Study to Assess the Bioequivalence of Trastuzumab Via Different Subcutaneous Delivery Platforms in Healthy Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP44770
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants will receive formulation 1 of trastuzumab SC via OBDS or HHS/SP with IS.
  Interventions: Drug: Trastuzumab
- Part 2 (Experimental): Participants will receive formulation 2 of trastuzumab SC via OBDS or HHS/SP with IS.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered to participants as a solution for injection.

SUMMARY:
This two-part study will evaluate the bioequivalence, safety, and tolerability of a single SC dose of trastuzumab administered via handheld syringe/syringe pump (HHS/SP) with infusion set (IS) and an on-body delivery system (OBDS).

ELIGIBILITY:
Inclusion Criteria:

* Within body mass index (BMI) range 18 to 38 kilogram per meter square (kg/m2), inclusive. Body weight <=100 kg
* Left ventricular ejection fraction (LVEF) >= 55 percent (%) measured by echocardiogram (ECHO)
* Negative test result for drugs of abuse
* Negative test result for hepatitis B surface antigen, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody screen
* Negative test for latent Tuberculosis (TB) infection by QuantiFERON® TB Gold
* Agree to use contraception and will refrain from sperm donation

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, respiratory, gastrointestinal, immunological, neurological, or psychiatric disorder; acute infection; or other unstable medical disease
* History of moderate or severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins
* Known sensitivity to recombinant hyaluronidase or other form of hyaluronidase
* History or presence of atrial fibrillation
* History of any clinically significant or clinically relevant cardiac condition
* History or presence of clinically significant electrocardiogram (ECG) abnormalities
* History of uncontrolled hypertension, hyperlipidemia, thyroid disorder, or diabetes
* Family history of clinically significant and clinically relevant hypersensitivity, allergy, or severe cardiac diseases
* History of previous anti-cancer treatments including pertuzumab, trastuzumab, anthracyclines, or any cardiotoxic drugs
* History of active or latent TB, regardless of treatment history
* Poor peripheral venous access
* History or presence of any malignancy, with the exception of completely excised basal cell or squamous cell carcinoma of the skin

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 312 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: Area Under the Concentration-Time Curve from Hour 0 to 21 days Postdose (AUC0-21days) of Trastuzumab | Up to Day 57
Part 1: Maximum Observed Concentration (Cmax) of Trastuzumab | Up to Day 57
Part 2: AUC0-21days of Trastuzumab | Up to Day 57
Part 2: Cmax of Trastuzumab | Up to Day 57
Percentage of Participants with Adverse Events (AEs) | Up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - Daytona Beach Clinical Rsch Unit, Daytona Beach, Florida
  - QPS Bio-Kinetic, Springfield, Missouri
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No